CLINICAL TRIAL: NCT03858959
Title: A Topical Desiccant Agent in Association With Manual Debridement in the Initial Treatment of Peri-implant Mucositis: a Clinical and Microbiological Pilot Study
Brief Title: A Topical Desiccant Agent in Association With Manual Debridement in the Treatment of Peri-implant Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Giorgio Lombardo, Associate Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UVerona
Record Dates: First submitted 2019-02-25; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HYBENX® Oral Tissue decontaminantTM (HBX) (Experimental): HYBENX® Oral Tissue decontaminantTM is a concentrated aqueous solution of sulfonated aromatics and free sulphates. Once placed onto susceptible organic material, the product instantly absorbs free and electrostatically bonded water, denaturing the molecular structure of the organic matter. Biofilm is expected to be especially sensitive to the disruptive action of HBX solution by virtue of its porous structure and high water content.
  Interventions: Device: topical agent
- Chlorhexidine Digluconate CorsodylTM (CHX) (Active Comparator): Chlorhexidine Digluconate CorsodylTM Dental Gel 1% is an antiseptic gel with cationic nature, effective against a wide range of Gram positive and negative bacteria, favourable to the plaque control and oral inflammation prevention.
  Interventions: Device: topical agent

INTERVENTIONS:
Device: topical agent — HBX protocol consisted in product application into the periodontal pocket (starting from the base) with a delivery syringe, second saline solution irrigation after 60 seconds to flush-out the product and Teflon-curettes debridement to remove the deposits.
  CHX protocol consisted in Teflon-curettes debridement to remove the deposits, associated with a first saline solution irrigation, and product application into the periodontal pocket (starting from the base) with a delivery syringe.

SUMMARY:
In patients presenting peri-implant mucositis, effective sub-mucosal debridement is crucial to prevent peri-implantitis. The aim of this pilot study was to assess the 3-month clinical and microbiological effects of a locally delivered liquid desiccant agent with molecular hygroscopic properties, in association with sub-gingival manual debridement, in sites with peri-implant mucositis.

Twenty-three patients presenting at least one implant with no radiographically detectable bone loss, a pocket probing depth ≥ 4 mm and bleeding on probing, were included in a 3-month randomized, parallel-groups, single-blind, prospective study. At baseline (T0), patients were randomly assigned to receive a desiccant liquid agent with molecular hygroscopic properties before debridement (Test-Group), or a Chlorhexidine 1% disinfectant gel after debridement (Control-Group). Treatments were performed also after 7 and 14 days. Peri- implant soft tissues assessment (PPD, BOP, mBI, VPI, mPLI) and microbial sampling were assessed at baseline and at 3-month follow-up (T1).

DETAILED DESCRIPTION:
A single-center, single-masked, parallel-groups, randomized clinical and microbiological study, was conducted between July and October 2018 at the Dentistry and Maxillo-facial Surgery Clinic, Department of Surgery, Dentistry, Paediatrics and Gynaecology (DIPSCOMI), University of Verona, Verona, Italy. The experimental protocol (Protocol HX-GL-ITA13, approval date 20/11/2013) was approved by the Ethical Committee of the University of Verona. The study was conducted in accordance with the Ethical Principles of the 64th World Medical Association Declaration of Helsinki and was consistent with good clinical practices. All participants signed a written informed consent.

The subjects were enrolled among individuals examined through a survey on prevalence of peri- implant infections (mucositis and peri-implantitis) in single-crown plateau-design locking-taper implants with a 3-year follow-up period. Twenty-three patients, aged between 37 and 71 years, met the study criteria.

Patients were randomly assigned (using a predefined computer-generated randomization scheme) to the Test-Group, which received the administration of a desiccant liquid with molecular hygroscopic properties (HYBENX® Oral Tissue decontaminantTM, HBX) before SRP, or to the Control-Group, which received the administration of a disinfectant gel after SRP (Chlorhexidine Digluconate CorsodylTM Dental Gel 1%, CHX).

Chlorhexidine Digluconate CorsodylTM Dental Gel 1% is an antiseptic gel with cationic nature, effective against a wide range of Gram positive and negative bacteria, favourable to the plaque control and oral inflammation prevention. HYBENX® Oral Tissue decontaminantTM is a concentrated aqueous solution of sulfonated aromatics and free sulphates. Once placed onto susceptible organic material, the product instantly absorbs free and electrostatically bonded water, denaturing the molecular structure of the organic matter. Biofilm is expected to be especially sensitive to the disruptive action of HBX solution by virtue of its porous structure and high water content. On the Test-Group of this study, HBX was administered before the Teflon-curettes debridement and left in contact with supra and sub-gingival plaque biofilm for up to 60 seconds, then rinsed with water and evacuated.

At baseline (T0) subjects were randomly assigned to the Test-Group or to the Control-Group, in order to be examined for microbial sampling, peri-implant soft tissues assessment and radiographic bone levels. The implants were consequently treated with HBX, before a SRP professional session, or CHX, after a SRP professional session. The treatment, performed by the same operator, was then repeated on days 7 and 14.

ELIGIBILITY:
Inclusion Criteria:

- presence of at least one implant with a pocket probing depth (PPD) ≥ 4 mm, bleeding on probing (BOP) or pus on probing and no radiographically detectable bone loss (Qualifying site).

Exclusion Criteria:

* pregnant or lactating females;
* patients with severe systemic diseases, or with uncontrolled diabetes mellitus;
* assumption of agents affecting the periodontal status within 1 month prior to the study;
* use of systemic antibiotics within 3 months prior to the study;
* prophylactic antibiotics requirement;
* peri-implant specific treatments within 6 months prior to the study;
* allergy to sulphates and its derivatives.

Ages: 37 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth (PPD) | 2 minutes
  PPD is recorded in mm as the distance between the gingival margin and the base of the periodontal pocket. The possible scale range is from 1 to 10 mm. The higher is the measure, the worst is the value. The measure is assessed at baseline (T0) and at 3-month recall appointment (T1) using a periodontal probe (Florida Probe; Florida Probes Company, Gainesville, FL, US), applying a force of mild intensity on each of the six sites of the implant, three (mesial, central, distal) on the buccal side and three on the lingual/palatal side.
Bleeding on probing (BOP) | 2 minutes
  BOP is recorded as 0 (no bleeding) or 1 (yes bleeding) after probing. It is a dichotomous dimensionless index with two possible values (0 and 1). It is assessed at baseline (T0) and at 3-month recall appointment (T1) using a periodontal probe (Florida Probe; Florida Probes Company, Gainesville, FL, US), applying a force of mild intensity on each of the six sites of the implant, three (mesial, central, distal) on the buccal side and three on the lingual/palatal side.
Modified Bleeding Index (mBI) | 2 minutes
  mBI is recorded as 0, 1, 2, 3 according to Mombelli et al. It is a dimensionless index with four possible values and a scale range from 0 to 3 (3 is the most abundant bleeding and the worst value). It is assessed at baseline (T0) and at 3-month recall appointment (T1) using a periodontal probe (Florida Probe; Florida Probes Company, Gainesville, FL, US), applying a force of mild intensity on each of the six sites of the implant, three (mesial, central, distal) on the buccal side and three on the lingual/palatal side.
Modified Plaque Index (mPLI) | 2 minutes
  mPLI is recorded as 0, 1, 2, 3 according to Mombelli et al. It is a dimensionless index with four possible values and a scale range from 0 to 3 (3 is the most abundant plaque and the worst value). It is assessed at baseline (T0) and at 3-month recall appointment (T1) using a periodontal probe (Florida Probe; Florida Probes Company, Gainesville, FL, US), applying a force of mild intensity on each of the six sites of the implant, three (mesial, central, distal) on the buccal side and three on the lingual/palatal side.
Visible Plaque Index (VPI) | 2 minutes
  VPI is recorded as 0 (no plaque) or 1 (yes plaque) after probing. It is a dichotomous dimensionless index with two possible values (0 and 1). It is assessed at baseline (T0) and at 3-month recall appointment (T1) using a periodontal probe (Florida Probe; Florida Probes Company, Gainesville, FL, US), applying a force of mild intensity on each of the six sites of the implant, three (mesial, central, distal) on the buccal side and three on the lingual/palatal side.

SECONDARY OUTCOMES:
Bacterial count (aerobic and anaerobic) | 3 days
  The concentration of bacteria in the plaque is expressed as CFU / mg of plaque. After supra-gingival plaque removal, the deepest site was isolated with sterile cotton rolls in order to properly collect a plaque sample (1 mg ca), through two paper points inserted and left for 30 seconds at the base of the periodontal pocket. The collected plaque sample was put in an Eppendorf tube containing thioglycolate medium (BD Difco) for cultural investigations.Plates were incubated at 37°C for 48 hours under specific conditions (Columbia blood agar and Schaedler blood agar). Colonies that appeared were counted and results refer to CFU/mg (colony-forming units per mg of plaque).

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Lombardo, Principal Investigator — Università di Verona
Locations (1):
- Giorgio Lombardo, Verona, Italy

IPD SHARING:
Plan to Share IPD: No